CLINICAL TRIAL: NCT00066963
Title: Comprehensive Oral Health Center for Discovery: New Strategies for Enhancing Tissue Integrity and Repair Early Childhood Caries: Prevention and Treatment Outcomes
Brief Title: Fluoride Varnish Randomized Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NIDCR-13058
Record Dates: First submitted 2003-08-07; First posted 2003-08-08 (Estimated); Results first posted 2012-05-08 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Dental Caries
Keywords: Early Childhood Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Counseling Only (No Intervention): Counseling Only
- FV every 12mo for 24mo + Counsel (Experimental): Preventive fluoride varnish every 12mo for 24mo plus Counseling
  Interventions: Device: Fluoride Varnish
- FV every 6mo for 24mo + Counseling (Experimental): Preventive fluoride varnish every 6mo for 24mo plus Counseling
  Interventions: Device: Fluoride Varnish

INTERVENTIONS:
Device: Fluoride Varnish — 0.1 mL (1 drop) applied on each of 2 arches
  Other Names: Duraphat® (Colgate Oral Pharmaceuticals)
  Arms: FV every 12mo for 24mo + Counsel; FV every 6mo for 24mo + Counseling

SUMMARY:
The purpose of this study is to compare the efficacy of fluoride varnish (FV) applied once or twice a year with counseling to counseling alone in preventing early childhood caries (ECC) (tooth decay in children under the age of five).

DETAILED DESCRIPTION:
This project was a prospective, randomized clinical trial (RCT) among initially caries-free children from about six months old (when primary teeth erupt) up to age three at two public health facilities in San Francisco, one serving a primarily Latino and one a primarily Asian population. The RCT 1) Compared the efficacy of once or twice/year fluoride varnish (FV) application and counseling to counseling alone in preventing early childhood caries (ECC); 2) Assessed pre-intervention salivary markers (biologic and chemical), behavioral and demographic factors as predictors of ECC; 3) Compared the efficacy of these interventions between sites serving different ethnic populations with a high prevalence of ECC; and 4) Determined the salivary fluoride release profile following exposure to fluoride varnish.

ELIGIBILITY:
Inclusion

* Children < 44 months old
* Caries-free
* 4 erupted maxillary incisors
* Residing in fluoridated community (San Francisco)

Exclusion

* Cleft Palate
* Developmental or learning disabilities
* Children with transient residence (homeless, migrant, foster home)
* Children with an another household member participating in the study

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 376 (Actual)
Dates: Start 2002-10; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane A Weintraub, DDS, MPH, Principal Investigator — University of California, San Francisco (now Univ North Carolina); Francisco Ramos-Gomez, DDS, MPH, Study Director — University of California, San Francisco (now Univ Calif Los Angeles)
Locations (1):
- UCSF School of Dentistry, San Francisco, California, United States

REFERENCES:
- [Result] Weintraub JA, Ramos-Gomez F, Jue B, Shain S, Hoover CI, Featherstone JD, Gansky SA. Fluoride varnish efficacy in preventing early childhood caries. J Dent Res. 2006 Feb;85(2):172-6. doi: 10.1177/154405910608500211. PMID 16434737
- [Result] Gansky SA, Cheng NF, Koch GG. Dose-Weighted Adjusted Mantel-Haenszel Tests for Numeric Scaled Strata in a Randomized Trial. Stat Biopharm Res. 2011 May 1;3(2):266-275. doi: 10.1198/sbr.2011.10014. PMID 21709814
- [Result] Lazar AA, Gansky SA, Halstead DD, Slajs A, Weintraub JA. Improving Patient Care Using the Johnson-Neyman Analysis of Heterogeneity of Treatment Effects According to Individuals' Baseline Characteristics. J Dent Oral Craniofac Epidemiol. 2013 Oct 1;1(3):19-33. PMID 25705704

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2001 - July 2002. Supplemental Nutrition Program for Women, Infants & Children (WICs); Womens resource center; medical clinics; pre-schools; dental clinics
Pre-assignment Details: Cleft lip or palate, developmental or learning disabilities, older than 36 mos; younger than 6 mos,immuno-compromised, born outside SF Bay Area where water is non-fluoridated, lack parental consent; lack 4 maxillary incisors, have caries, other family member in study, transient parents, ineligible to use SF Health Dept service
Groups:
- No Intervention: Counseling Only: Counseling Only (0FV)
- Experimental: FV Every 12mo for 24mo + Counsel: Preventive fluoride varnish every 12mo for 24mo plus Counseling (2FV)
- Experimental: FV Every 6mo for 24mo + Counsel: Preventive fluoride varnish every 6mo for 24mo plus Counseling (4FV)
Period: Overall Study
Arm/Group | No Intervention: Counseling Only | Experimental: FV Every 12mo for 24mo + Counsel | Experimental: FV Every 6mo for 24mo + Counsel
Started | 126 | 124 | 126
Completed | 100 (any follow-up) | 93 | 87
Not Completed | 26 | 31 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Intervention: Counseling Only | Experimental: FV Every 12mo for 24mo + Counsel | Experimental: FV Every 6mo for 24mo + Counsel | Total
Number analyzed (Participants) | 126 | 124 | 126 | 376
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 126 | 124 | 126 | 376
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Year] | 1.8 (0.6) | 1.8 (0.5) | 1.8 (0.6) | 1.8 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 66 | 64 | 198
  Male | 58 | 58 | 62 | 178
Region of Enrollment [Number; unit: participants]
  United States | 126 | 124 | 126 | 376

OUTCOME MEASURES:

1. Primary Outcome: Number of Caries Incident Cases
Description: A trained, calibrated dentist blinded to treatment arm performed visual-tactile dental exams at 1 and 2 years post-baseline. Group-specific number of incident cases were reported as the number of individual participants with caries at a follow-up visit.
Time Frame: two years
Population: intention-to-treat with any follow-up information. multiple imputation for sensitivity analyses.
Measure: Number; unit: participants
Groups:
- Counseling Only: caregiver counseling only (zero fluoride varnish)
- FV 1x/Year + Counseling: fluoride varnish (FV) (5% NaF, Duraphat®, Colgate) once per year for 2 years (every 12 months) plus caregiver counseling
- FV 2x/Year + Counseling: fluoride varnish (FV) (5% NaF, Duraphat®, Colgate) twice per year for 2 years (every 6 months)
Arm/Group | Counseling Only | FV 1x/Year + Counseling | FV 2x/Year + Counseling
Number analyzed (Participants) | 100 | 93 | 87
participants | 42 | 23 | 14
Statistical Analysis 1: Comparison: Counseling Only vs FV 1x/Year + Counseling vs FV 2x/Year + Counseling; Planned sample size of 384 participants (128/study arm) (alpha = 0.05, power = 90%, 50% attrition, χ2 test) to detect caries incidence differences, based on caries incidence in the literature (20% to 50% over two years). 50% attrition in the sample size calculation was selected based on the literature (e.g. Weinstein et al., 1994 reported 53% attrition in six months.); Test type: Superiority or Other; p < 0.001, Mantel Haenszel; 2 d.f; Odds Ratio (OR) = 3.8, 95% CI 2-sided [1.9 to 7.6] — Counseling Only vs FV 2x/yr+Counseling

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | No Intervention: Counseling Only | Experimental: FV Every 12mo for 24mo + Counsel | Experimental: FV Every 6mo for 24mo + Counsel
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/93 | 0/87
Other Adverse Events (participants affected / at risk) | 0/100 | 0/93 | 1/87
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Intervention: Counseling Only (N=100) | Experimental: FV Every 12mo for 24mo + Counsel (N=93) | Experimental: FV Every 6mo for 24mo + Counsel (N=87)
Ulcer on the cheek (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Upon questioning, a parent reported at the 18-month visit the child had an "ulcer on the cheek" onsetting 2 months after the last fluoride varnish application, which was a "fluoride-free" placebo application. The ulcer was gone at the 24-month visit.

LIMITATIONS AND CAVEATS:
In a protocol deviation, children received placebo varnish for 10 months; this would be expected to bias the study toward the null of no difference among groups. The study did not address FV efficacy for children with extant or past caries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No